CLINICAL TRIAL: NCT06578975
Title: HT-ENDO: A Multiomics-based Biomarker for the Diagnosis of Endocrine Hypertension: a Pragmatic, Diagnostic, Randomized, Outcome-based Trial
Acronym: HT-ENDO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: JDeinum (Other)
Responsible Party: Sponsor-Investigator, JDeinum, Principal Investigator, Radboud University Medical Center
Organization: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 115632
Record Dates: First submitted 2024-03-11; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-Omics diagnosis (Experimental): Participants in this arm will be diagnosed with the mutli-omics based biomarker
  Interventions: Diagnostic Test: HT-ENDO-MOS-A13
- Normal diagnosis (Other)
  Interventions: Other: Normal diagnosis

INTERVENTIONS:
Diagnostic Test: HT-ENDO-MOS-A13 — Mutli-Omics based biomarker to diagnose primary hypertension or endocrine forms of hypertension; primary aldosteronism, pheochromocytoma/functional paraganglioma or Cushing syndrome.
  Arms: Multi-Omics diagnosis
Other: Normal diagnosis — Standard diagnosis for endocrine hypertension
  Arms: Normal diagnosis

SUMMARY:
Rationale: Diagnosis of endocrine forms of hypertension (primary aldosteronism, pheochromocytoma/paraganglioma and Cushing syndrome) is a lengthy and tedious process. Recently a multiomics biomarker was developed through machine learning that shows high accuracy in predicting the presence of endocrine hypertension or primary hypertension. Given the propensity to data shift in applications of machine learning derived algorithms validation of this multiomics biomarker in a prospective comparative trial is warranted.

Objective: To determine the diagnostic performance of the new diagnostic biomarker

Study design: A randomized, diagnostic, outcome-based trial

Study population: Hypertensive patients 18-75 yrs, referred to ESH Hypertension Excellence centers, who may suffer from endocrine hypertension.

Intervention (if applicable): One group is diagnosed by classic endocrine tests, the other by the multiomics biomarker. Ensuing treatment depends on diagnosis and subtyping results.

Main study parameters/endpoints:

Primary endpoint is potency of antihypertensive medication to reach a target systolic blood pressure value of 135 mm Hg by home blood pressure measurement or an equivalent value for ambulatory blood pressure measurement, standardized office blood pressure measurement or unattended automatic blood pressure measurement.

Secondary endpoints: Ambulatory blood pressure, biochemical cure of endocrine hypertension (if treated by surgery), costs, quality of life

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: In the control group patients follow the same diagnostic itinerary as in usual care. In the biomarker group, endocrine tests will have been replaced by a blood and urine collection. The risk in both arms consists of missing an endocrine diagnosis. From the preceding accuracy study this risk is low for the use of the biomarker. After 6 months follow-up patients that were diagnosed by the biomarker may switch to a classic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Have a properly documented hypertension by abpm, hbpm, unattended office blood pressure measurement or carefully performed office measurement.
* Has a physician who feels an urge to exclude or diagnose EHT for one or more of the following reasons
* resistant hypertension AND/OR
* hypokalemia, spontaneous or diuretic-induced AND/OR
* history or physical examination suggestive of endocrine hypertension
* Willingness and ability to give informed consent

Exclusion Criteria:

* White-coat hypertension
* Known renal artery stenosis
* Known licorice abuse
* Known familial form of endocrine hypertension
* Cardiovascular event (myocardial infarction, cerebrovascular event) < 6 months [Y/N]
* Hypertensive crisis < 6 months
* eGFR < 50 ml/min/1,73m2
* Liver failure
* Known severe valvular or structural heart disease (excluding left ventricular hypertrophy)
* NYHA class III or IV heart failure or known reduced left ventricular function (ejection fraction (EF) <30%)
* EKG demonstrating significant pathology (e.g. myocardial infarction, atrial fibrillation, or any other cardial condition prohibiting start of study medication)
* Life expancy < 1 year
* For women, current pregnancy or unprotected intercourse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Potency of antihypertensive medication | from date of start of treament until end of study evaluation (6 months)
  Primary endpoint is potency of antihypertensive medication to reach a target systolic blood pressure value of 135 mm Hg by home blood pressure measurement or an equivalent value for ambulatory blood pressure measurement, standardized office blood pressure measurement or unattended automatic blood pressure measurement.

SECONDARY OUTCOMES:
Ambulatory blood pressure | from date of start of treament until end of study evaluation (6 months)
  Ambulatory blood pressure decrease comparison of the two diagnostic methods
Biochemical cure of endocrine hypertension (if treated by surgery) | from date of start of treament until end of study evaluation (6 months)
  Comparison of effectiveness of biochemical cure of endocrine hypertension (if treated by surgery) As defined by normalisation of aldosterone and renin levels in case of adrenalectomy for aldosterne producing adenoma, normalization of (nor)metanephrine levels after surgery for pheochromocytoma, or normalization of cortisol levels after hypophysectomy or adrenalectomy in Cushing disease/syndrome.
Cost | from date of randomization until end of study evaluation (6 months)
  Cost-effectiveness comparison between the two diagnostic methods.for a cost-effectiveness analysis we will use the costs of all procedures and the results of the EQ-5D questionnaire.
Quality of life EQ-5D (min 00000- max 55555, with 55555 having the best quality of life) | from date of start of treament until end of study evaluation (6 months)
  Quality of life comparison between participants in the two arms using the EQ-5D
Quality of life SF-36 (36-Item Short Form Health Survey, 0-100 for each scale, lower means worse qulaity of life) | from date of start of treament until end of study evaluation (6 months)
  Quality of life comparison between participants in the two arms using the SF-36

OTHER OUTCOMES:
Extra standard analysis | From end of follow-up of trial to initial diagnosis confirmed or not (around 3 months)
  proportion of participants diagnosed with PHT in the intervention MOMICS-ENDO arm who choose to undergo a standard analysis after the end of follow-up
EHT after secondary standard analysis | From end of follow-up of trial to initial diagnosis confirmed or not (around 3 months)
  number of participants with PHT in the MOMICS-ENDO arm who have EHT after a secondary standard analysis after the end of follow-up.
carbon footprints of both arms | from inclusion to end of follow-up (6 months after start of treatment)
  comparison of the carbon footprints of both arms

IPD SHARING:
Plan to Share IPD: Undecided